CLINICAL TRIAL: NCT03509428
Title: A Pragmatic Factorial Design Randomised Controlled Study to Assess the Efficacy of the Implementation of a Prehabilitation Programme in Patients Undergoing Elective Major Intra - Cavity Cancer Surgery in Wessex
Brief Title: The Wessex Fit-4-Cancer Surgery Trial
Acronym: WesFit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Portsmouth Hospitals NHS Trust (Other Government); Hampshire Hospitals NHS Foundation Trust (Other); Poole Hospital NHS Foundation Trust (Other); Isle of Wight NHS Trust (Other); Dorset County Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RHM CRI 0360
Record Dates: First submitted 2018-03-07; First posted 2018-04-26 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Exercise; mortality; morbidity; surgery; colorectal; upper gastrointestinal; hepatobiliary; urology; lung; nutrition; psychology
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design randomised controlled interventional trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking of CPET assessors and dual reporting, masking of personnel involved in outcome data collection, masking of sarcopenia assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Usual care plus additional monitoring
- SRETP (Experimental): Structured Responsive Exercise Training Programme (SRETP) prior to surgery
  Interventions: Behavioral: SRETP
- Psychological support (Experimental): Psychological support prior to surgery
  Interventions: Behavioral: Psychological support
- SRETP and psychological support (Experimental): Structured Responsive Exercise Training Programme (SRETP) and psychological support prior to surgery
  Interventions: Behavioral: SRETP; Behavioral: Psychological support

INTERVENTIONS:
Behavioral: SRETP — SRETP will involve short periods of exercise at a high intensity interspersed with short periods of exercise at a moderate intensity (aerobic interval training). We will also include resistance training in each session. Exercise intensities during the interval exercise-training program are specific to each patient and derived from CPET. Moderate intensity exercise is below the anaerobic threshold (AT). Patients will exercise at 80% of oxygen uptake (VO2) obtained at the anaerobic threshold (80%AT) for moderate intensity exercise - 3 minutes. Severe exercise intensity is recognised as 50% of the difference between the VO2 AT and VO2 Peak (50%∆) - 2 minutes.
  Arms: SRETP; SRETP and psychological support
Behavioral: Psychological support — Support sessions will be patient-centred, giving the patient an opportunity to raise any issues/concerns they are having, this may include (but will not be limited to) ways of coping with their reactions to cancer, family and relationship issues, exploring personal issues and dealing with practical issues. Patients will have access to other resources available at the cancer centres including but not restricted to further information about their condition and how to access financial support. These processes reflect the best practice currently being delivered by cancer support centre staff in the Wessex region. Any patient deemed at risk (i.e. from suicidal ideation or self harm) will be reported to their GP, followed up by a letter.
  Arms: Psychological support; SRETP and psychological support

SUMMARY:
Trial Phase: Phase III: A multi-centre efficacy pragmatic factorial design randomised controlled trial with patient informed development and process evaluation

Indication: Patients undergoing major electively resectable intra - cavity cancer surgery with or without neoadjuvant cancer treatments (including chemotherapy (NAC), chemoradiotherapy (CRT), or immunotherapy).

Objective: To investigate the efficacy of a community based Structured Responsive Exercise-training Programme (SRETP) ± psychological support on surgical outcome by reducing postoperative length of stay (LOS) and complications.

Secondary Objective:

To investigate the efficacy of a community based Structured Responsive Exercise-training Programme (SRETP) ± psychological support to improve disease-free overall survival. Cardiopulmonary Exercise test (CPET) variables, physical activity, morbidity, radiological markers of sarcopenia, toxicity, tumour down-staging, tumour regression, disability adjusted survival (WHODAS) overall survival and quality of life (QoL).

DETAILED DESCRIPTION:
Rationale: Fitter patients have better surgical outcomes. Poor physical fitness measured objectively using cardiopulmonary exercise testing has been associated with increased LOS, increased morbidity and mortality in many patient cohorts undergoing major cancer surgery. Chemotherapy and radiotherapy have detrimental effects on physical fitness, which may in turn have a detrimental effect on the patients' ability to withstand surgery. Research suggests psychological factors including depression and self-efficacy (confidence to manage cancer-related problems) prior to surgery predict recovery trajectories in health-related quality of life up to 2 years after major surgery for colorectal cancer.

The aim is to investigate whether SRETP (Prehabilitation) ± psychological support prior to and during cancer treatment before major elective surgery reduces LOS, increases survival and improves their ability to self manage. Additionally, we aim to see if this intervention can bring about long-term behavioural change in relation to physical activity.

Trial Design: Phase III: A pragmatic factorial design randomised controlled to assess the effectiveness of a prehabilitation programme delivered prior to cancer treatments and/or major cancer surgery in patients undergoing elective intra-cavity major cancer surgery in Wessex.

Sample size: 1560

Intervention:

1. An in-hospital transition to a community based Structured Responsive Exercise-Training Programme (SRETP) ± psychological support (delivered in community/ council gyms or Cancer Support Centers). The intervention/s will be delivered before surgery. Patients receiving neoadjuvant cancer treatments prior to surgery will receive the intervention during and after these treatments.
2. Control: Standard care with extra monitoring

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* aged over 18 years old
* scheduled to have major intra-cavity cancer surgery with a curative intent, defined as thoracic, colorectal, oesophagogastric, urological and hepatobiliary (inc. pancreatic).
* surgery alone (unimodal)
* surgery combined (multimodal) with cancer treatments (neoadjuvant chemotherapy, chemoradiotherapy or immunotherapies).
* All patients deemed by the MDT as potentially curable or undergoing neoadjuvant cancer treatments prior to restaging and surgery.

Exclusion Criteria:

* Patients will be excluded if under the age of 18 years,
* if their tumour is considered surgically non- resectable,
* having absolute or relative contraindications to completing a CPET,
* patients are unable to perform CPET due to other coexisting acute illness or conditions (e.g. lower limb dysfunction),
* patients decline surgery,
* if their weight exceeds 145kg
* patients unable to give informed consent.
* Patients having >2 mm ST depression if symptomatic or 4 mm if asymptomatic or >1 mm ST elevation during any CPET will need to be withdrawn from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative length of hospital stay | up to 1 year
  Date of hospital admission minus date of discharge would equal length of post-operative stay (LOS).

SECONDARY OUTCOMES:
Change in objectively measured cardiopulmonary exercise testing variables - Oxygen uptake at anaerobic threshold (ml/kg/min) and oxygen uptake at peak exercise (ml/kg/min) | up to 15 weeks
  Change in cardiopulmonary exercise variables i.e. oxygen uptake (VO2) at anaerobic threshold (AT) and at peak exercise. A clinically significant difference in physical fitness is defined as ≥ 2ml/min/kg VO2 at AT.
Overall survival - 1 | 1 year post-operatively
  Overall survival at 1 year post surgery
Overall survival -2 | 5 years post-operatively
  Overall survival at 5 year post surgery
Disease free survival | 1 year post-operatively
  Clinical or radiologically measured disease free survival
Post-operative morbidity -1 | POMS at day 3,5,7 and 15.
  Patients post-operative morbidity survey (POMS) will be characterised on day 3, 5, 7 and 15. The POMS 18-item survey will be used to address nine domains of postoperative morbidity (pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, wound complication, haematological and pain).
Post-operative morbidity -2 | up to 1 year
  On day of discharge, patient's surgical complications (if any) will be graded using the Clavien-Dindo classification of surgical complications This classification is used to assess overall hospital morbidity following surgical procedures. Patients are graded as 0 (no complications) or Grade I-V based on the level of complication, including the number of organ system involvement. Grade V is defined as death of a patient. A record of the Comprehensive Complication Index (CCI) - an update of the Clavien-Dindo classification will also be collected
Physical activity -1 | Baseline up to 1 year post-operatively
  Number of steps while active using a triaxial accelerometer eg. Senseware
Physical activity -2 | Baseline up to 1 year post-operatively
  sleep efficiency using a triaxial accelerometer eg. Senseware
Physical activity -3 | Baseline up to 1 year post-operatively
  metabolic equivalents using a triaxial accelerometer eg. Senseware
Physical activity -4 | Baseline up to 1 year post-operatively
  Godin Leisure Time and Exercise questionnaire - A self-reported measure of physical activity
Health related quality of life -1 | Baseline up to 1 year post-operatively
  Changes in health related quality of life measurements using validated questionnaires; including:
  EQ-5D-5L is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys
Health related quality of life -2 | Baseline up to 1 year post-operatively
  Changes in health related quality of life measurements using validated questionnaires; including:
  Cancer specific quality of life will be measured using the EORTC-QLQ-C30.
Health related quality of life -3 | Baseline up to 1 year post-operatively
  Changes in health related quality of life measurements using validated semi-structured interview techniques
Mental well being -1 | Baseline up to 1 year post-operatively
  Self-efficacy (confidence) to self-manage chronic disease (SEMCD), measured using the Lorig SEMCD scale
  A confidence scale that represents the patients confidence that a regular task can be achieved. 1 = Not confident at all and 10= totally confident.
Mental well being -2 | Baseline up to 1 year post-operatively
  Patients knowledge skills and confidence to manage their own health and care will be measured using the Patient Activation Measure (PAM)
  Agreement or disagreement with statements. Choice between disagree strongly, disagree, agree, agree strongly and not applicable
Mental well being -3 | Baseline up to 1 year post-operatively
  Anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS)
  A tick box questionnaire relating to anxieties and depression that a patient might have felt over the past week. Choices are most of the time, a lot fo the time, from time to time, and not at all for most questions.
Mental well being -4 | Baseline up to 1 year post-operatively
  Resilience, measured using the Connor-Davidson Resilience Scale (CD-RISC2)
  Patients are asked to choose "x" in a box that best indicates how much they agree with the following statements resilience over the past month.
  Options are not at all true; rarely true; sometimes true; often true; true nearly all of the time
Mental well being -5 | Baseline up to 1 year post-operatively
  Brief illness perception questionnaire (B-IPQ) - A self- reported nine-item scale designed to rapidly assess the cognitive and emotional representations of illness by a questionnaire.
  Various illness questions are asked and the patient picks a number from 0 to 10; 0= no affect at all and 10= severely affects my life.
Complex health interventions evaluation | Baseline up to 1 year post-operatively
  Medical research council (MRC) RE-AIM reporting
Radiological markers of sarco-cachexia measured from routine CT scans | Baseline up to 1 year post-operatively
  CT, MRI, PET CT full report from radiologist including TNM stage, venous invasion, resection margin involvement, tumour metabolic activity, RECIST staging and any other cancer pathway specific staging/restaging test. Raw DICOM files from radiological softwares or via the PACS team will be downloaded securely to measure radiological markers of sarco-cachexia.
Toxicity and adverse events | Baseline up to 1 year post-operatively
  Neoadjuvant cancer therapy induced toxicity measured using the CTC AE v4
Tumour outcomes -1 | Baseline up to 1 year post-operatively
  Radiology - CT, MRI, PET CT - Tumour Node Metastasis (TNM v7) stage
Tumour outcomes -2 | Baseline up to 1 year post-operatively
  Radiology - CT, MRI, PET CT full report from radiologist mainly including venous invasion
Tumour outcomes -3 | Baseline up to 1 year post-operatively
  Radiology - CT, MRI, PET CT full report from radiologist mainly including resection margin involvement
Tumour outcomes -4 | Baseline up to 1 year post-operatively
  Radiology - CT, MRI, PET CT full report from radiologist mainly including tumour metabolic activity
Tumour outcomes -5 | Baseline up to 1 year post-operatively
  Radiology - CT, MRI, PET CT full report from radiologist mainly including RECIST staging
Tumour outcomes -6 | Baseline up to 1 year post-operatively
  Radiology - CT, MRI, PET CT full report from radiologist mainly including tumour regression score
Tumour outcomes -7 | Baseline up to 1 year post-operatively
  Histopathology - TNM score version 7
Tumour outcomes -8 | Baseline up to 1 year post-operatively
  Histopathology - differentiation grading using TNM version 7
Tumour outcomes -9 | Baseline up to 1 year post-operatively
  Histopathology - extramural tumour extension using TNM version 7
Tumour outcomes -10 | Baseline up to 1 year post-operatively
  Histopathology - lymphovascular invasion using TNM version 7
Tumour outcomes -11 | Baseline up to 1 year post-operatively
  Histopathology - perineural invasion using TNM version 7
Tumour outcomes -12 | Baseline up to 1 year post-operatively
  Histopathology - venous invasion using TNM version 7
Tumour outcomes -13 | Baseline up to 1 year post-operatively
  Histopathology -resection margin status using TNM version 7
Tumour outcomes -14 | Baseline up to 1 year post-operatively
  Histopathology - tumour regression grading (TRG/ Mandard Score)
Tumour outcomes -15 | Baseline up to 1 year post-operatively
  Histopathology -lymph node status using TNM version 7
Tumour outcomes -16 | Baseline up to 1 year post-operatively
  Histopathology - number of lymph nodes involved using TNM version 7
Disability adjusted survival | Baseline up to 1 year post-operatively
  WHODAS v2.0 will ask patients to rate whether their health condition has had impact upon them in regards to 7 disability and functionality domains (understanding and communicating, getting around, self-care, getting along with others, life activities: household, life activities: work/school, and participation in society). This includes a measure of cost effectiveness.
Tumour microenvironment | Baseline up to 1 year post-operatively
  Endoscopic and surgical paired tumour biopsies will be taken as part of the oesophageal cancer clinical and molecular stratification study (OCCAMS) if the patient has been consented to the bio-banking study. Endoscopic and surgical paired tumour biopsies will be taken as part of TARGET LUNG study if the patient has been consented to the bio-banking study. Other tumor types will be banked in centers taking part in the International Cancer Genome Consortium. Clinical cancer pathway pathological samples embedded in paraffin and used in routine clinical practice may also be requested at a later stage for tumour analyses.
  Tumour biopsy +/- at endoscopic ultrasound (pre Cancer treatments and upon diagnosis) and at surgery (where possible depending on availability at site and cancer cohort)
Nutrition -1 | Baseline up to 1 year post-operatively
  Height (cms) and weight (kg) will be combined to report BMI in kg/m^2
Nutrition -2 | Baseline up to 1 year post-operatively
  Patient Reported Experience Measures (PREMS) including symptom and appetite questionnaires (Council of Nutrition Appetite Questionnaire- CNAQ) (in My Medical Record as part of standard clinical care)
Nutrition -3 | Baseline up to 1 year post-operatively
  Patient self-completing online assessment (myFood24 incorporated in My Medical Record)
Nutrition -4 | Baseline up to 1 year post-operatively
  Malnutrition Universal Screening Tool as part of standard clinical care

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Leggett, Study Director — University Hospitals Southampton NHS Foundation Trust
Locations (1):
- University Hopsitals Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] West M, Bates A, Grimmett C, Allen C, Green R, Hawkins L, Moyses H, Leggett S, Z H Levett D, Rickard S, Varkonyi-Sepp J, Williams F, Wootton S, Hayes M, P W Grocott M, Jack S. The Wessex Fit-4-Cancer Surgery Trial (WesFit): a protocol for a factorial-design, pragmatic randomised-controlled trial investigating the effects of a multi-modal prehabilitation programme in patients undergoing elective major intra-cavity cancer surgery. F1000Res. 2021 Sep 21;10:952. doi: 10.12688/f1000research.55324.2. eCollection 2021. PMID 36247802